CLINICAL TRIAL: NCT06132412
Title: Transcranial Direct Current Stimulation in Conjunction with Individualized Physical Therapy for Individuals with Chronic Knee Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Sangeetha Madhavan, Professor in Department of Physical Therapy, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-1323
Record Dates: First submitted 2023-10-30; First posted 2023-11-15 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Knee Pain Chronic
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active tDCS+PT (Experimental): For those participants assigned to the active or sham tDCS groups, the overall set-up will be identical between groups and will use the Mini-CT device. However, the sham tDCS group will have the tDCS device turned off after 30 seconds of stimulation. Saline-soaked sponge electrodes that are 35 cm^2 in size will be used for both the active and sham tDCS groups. For electrode placement, the active electrode (anode) will be placed over M1 contralateral to the side of primary knee pain (over C3/4 using the 10-20 system for electrode placement), while the reference electrode (cathode) will be over the contralateral supraorbital region, which is ipsilateral to the painful knee (Fp2 using the 10-20 system). The intensity will be set at 2mA for the active tDCS group, following a 30 second ramp-up time. The participants in the active tDCS group will undergo 20 minutes of tDCS treatment prior to receiving individualized PT intervention.
  Interventions: Device: transcranial direct current stimulation; Other: physical therapy
- sham tDCS+PT (Sham Comparator): For those participants assigned to the active or sham tDCS groups, the overall set-up will be identical between groups and will use the Mini-CT tDCS device. However, the sham tDCS group will have the tDCS device turned off after 30 seconds of stimulation. Saline-soaked sponge electrodes that are 35 cm^2 in size will be used for both the active and sham tDCS groups. For electrode placement, the active electrode (anode) will be placed over M1 contralateral to the side of primary knee pain (over C3/4 using the 10-20 system for electrode placement), while the reference electrode (cathode) will be over the contralateral supraorbital region, which is ipsilateral to the painful knee (Fp2 using the 10-20 system). The participants in the sham tDCS group will undergo 20 minutes of sham tDCS treatment prior to receiving individualized PT intervention.
  Interventions: Device: transcranial direct current stimulation; Other: physical therapy

INTERVENTIONS:
Device: transcranial direct current stimulation — Transcranial direct current stimulation (tDCS) is a form of noninvasive brain stimulation that can have neuromodulatory effects on central nervous system structures, specifically the primary motor cortex (M1), and can potentially target maladaptive plasticity and nociplastic sources of pain. There is both anodal and cathodal tDCS, anodal stimulation increases excitability of the cortex whereas cathodal stimulation decreases excitability. At the synaptic level, anodal tDCS induces effects that mimic long term potentiation (LTP), while cathodal tDCS results in long term depression.
  Other Names: tDCS
Other: physical therapy — Participants will receive individualized and impairment-based physical therapy treatment for their knee pain. This treatment can involve manual therapy, exercise or balance training depending on their particular needs.
  Other Names: PT

SUMMARY:
Background: There is a high prevalence of chronic pain in the US, with nearly half of adults experiencing chronic pain. Chronic pain is associated with impaired mobility, specifically ambulation. Treatment for chronic knee pain is complex given that pain is not only due to peripheral sources, but also due to alterations of the central nervous system (CNS). Majority of physical therapy (PT) interventions involve a bottom-up approach targeting the peripheral pain sources and many patients (~66%) do not respond to this treatment approach. Noninvasive brain stimulation techniques such as transcranial direct current stimulation (tDCS) is a novel and promising option for a top-down intervention that can have neuromodulatory effects on the CNS and may better target central factors associated with chronic pain. Purpose: To determine if tDCS delivered to the primary motor cortex in conjunction with individualized PT will result in greater improvements in pain and function compared to sham tDCS with individualized PT in individuals with chronic knee pain. Methods: This study will be performed at outpatient PT clinics at the University of Illinois Hospital. Eligible participants will include patients with chronic knee pain (duration > 3 months) who have not undergone surgery to this area and are scheduled to receive formal PT intervention. Subjects will be randomized to the active tDCS + PT group or sham tDCS + PT group and will receive the intervention for 8 sessions. Outcomes include pain ratings, pressure pain thresholds, patient specific functional scale, lower extremity functional scale, quadriceps strength, knee range of motion, 2-minute walk test, 5 time sit to stand, patient health questionnaire-2, and Central Sensitization Inventory. Impact: The use of adjuvant therapies such as tDCS have the potential to optimize rehabilitation treatment for individuals with chronic pain by offering a more comprehensive treatment that targets peripheral and central sources of pain.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years old
* Knee pain
* Knee pain duration >/= 3 months

Exclusion Criteria:

General exclusion criteria

* History of surgery on affected knee
* Pregnant

tDCS exclusion criteria

* Skin hypersensitivity
* History of contact dermatitis
* Any other skin or scalp condition that could be aggravated by tDCS
* Previous adverse reactions to tDCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment ratio | through study completion, an average of 1 year
  We will record the number of patients screened and enrolled in the study.
Pain (NPRS) | baseline, every follow-up session through study completion
  This will be measured subjectively using the Numeric Pain rating scale (NPRS). The PT or key research personnel with ask the participant their pain rating using a 0-10 scale. They will ask the current pain intensity rating, highest and lowest pain intensity rating in the past 2 week period.
Two-minute walk test (2MWT) | baseline, at final intervention session
  Distance walked, number of rest breaks and the assistive device(s) used during a 2MWT will be measured. From this test walking speed can also be calculated.

SECONDARY OUTCOMES:
Pressure pain threshold (PPT) | baseline, at final intervention session
  PPT will be obtained with an electronic pressure algometer and the pressure will be recorded in kPa to allow for comparison to norms
central sensitization inventory (CSI) | baseline, at final intervention session
  CSI is a self-report questionnaire that will be used as a secondary outcome to identify patients that may have symptoms related to central sensitization or nociplastic pain which may allow for subgroup analysis of data to occur
Lower extremity functional scale (LEFS) | baseline, at final intervention session
  self-report questionnaire where participants will rate the difficulty level they have with various daily mobility tasks
Patient specific functional scale (PSFS) | baseline, at final intervention session
  The PSFS is a self-report outcome measure that is individualized to the patient's specific activity impairments. The participant will choose 3 activities that are limited or difficult for them due to their knee pain and then will rate the level of difficulty of each task. On this scale, 0 means that the participant is unable to complete the activity at all and 10 means that the participant is able to perform the activity at the same level as before the injury or problem.
Five time sit to stand (5STS) | baseline, at final intervention session
  5STS will time the amount of time it takes for the participant to stand up and sit down five times as fast as they can from a standard chair without the use of their upper extremities if possible. If participants require upper extremity support to complete the task then this will be documented
knee range of motion (ROM) | baseline, at final intervention session
  ): Knee flexion and extension ROM will be measured with the patient in a supine position if possible. If participants have knee ROM measured in a position other than supine this will be documented.
quadriceps strength | baseline, at final intervention session
  Quadriceps strength will be assessed using a hand-held dynamometer with the patient in a seated position
Treatment adherence | through study completion, an average of 1 year
  Adherence to tDCS and physical therapy treatment will also be recorded.
tDCS satisfaction | at final intervention session
  Participants and clinicians involved in the study will also complete a survey following completion of the study regarding their impressions (positive and negative) regarding tDCS.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No